CLINICAL TRIAL: NCT00612040
Title: A 16 Week Randomised, Open Labelled, 3-armed, Treat-to-target, Parallel Group Trial Comparing SIBA (D) Once Daily + NovoRapid®, SIBA (E) Once Daily + NovoRapid® and Insulin Glargine Once Daily + NovoRapid®, All in a Basal/Bolus Regimen in Subjects With Type 1 Diabetes
Brief Title: Comparison of Two NN1250 Formulations Versus Insulin Glargine, All in Combination With Insulin Aspart in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-1835; 2007-002474-60 (EudraCT Number)
Record Dates: First submitted 2008-01-25; First posted 2008-02-11 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SIBA (D) (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- SIBA (E) (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- IGlar (Experimental)
  Interventions: Drug: insulin glargine; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Formulation 1: Treat-to-target dose titration scheme, injection s.c. (under the skin), once daily
  Arms: SIBA (D)
Drug: insulin degludec — Formulation 2: Treat-to-target dose titration scheme, injection s.c. (under the skin), once daily
  Arms: SIBA (E)
Drug: insulin glargine — Treat-to-target dose titration scheme, injection s.c., once daily
  Arms: IGlar
Drug: insulin aspart — Treat-to-target dose titration scheme, injection s.c. (under the skin), 3 times daily

SUMMARY:
This trial is conducted in Europe, Oceania and the United States of America (USA). The aim of this trial is to compare two NN1250 (insulin degludec) formulations with each other and with insulin glargine, all in combination with insulin aspart in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least one year
* HbA1c 7-11% (both inclusive)
* Treated with insulin for at least six months - any regimen

Exclusion Criteria:

* Any systemic treatment with products which in the Investigator's opinion could interfere with glucose or lipid metabolism (eg systemic corticosteroids) 3 months prior to randomisation
* Subject has a clinically significant, active (during the past 12 months) disease of the gastrointestinal, pulmonary, neurological, genitourinary, or haematological system that, in the opinion of the Investigator, may confound the results of the trial or pose additional risk in administering trial product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (30):
- United States (8):
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Renton, Washington
- Australia (5):
  - Novo Nordisk Investigational Site, Wollongong, New South Wales
  - Novo Nordisk Investigational Site, Keswick, South Australia
  - Novo Nordisk Investigational Site, East Ringwood, Victoria
  - Novo Nordisk Investigational Site, Geelong
  - Novo Nordisk Investigational Site, Miranda
- Germany (7):
  - Novo Nordisk Investigational Site, Aschaffenburg
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Saint Ingbert
- Norway (5):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Elverum
  - Novo Nordisk Investigational Site, Kristiansand
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
- Sweden (5):
  - Novo Nordisk Investigational Site, Alingsås
  - Novo Nordisk Investigational Site, Karlstad
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Umeå

REFERENCES:
- [Result] Birkeland KI, Home PD, Wendisch U, Ratner RE, Johansen T, Endahl LA, Lyby K, Jendle JH, Roberts AP, DeVries JH, Meneghini LF. Insulin degludec in type 1 diabetes: a randomized controlled trial of a new-generation ultra-long-acting insulin compared with insulin glargine. Diabetes Care. 2011 Mar;34(3):661-5. doi: 10.2337/dc10-1925. Epub 2011 Jan 26. PMID 21270174
- [Result] Home PD, Meneghini L, Wendisch U, Ratner RE, Johansen T, Christensen TE, Jendle J, Roberts AP, Birkeland KI. Improved health status with insulin degludec compared with insulin glargine in people with type 1 diabetes. Diabet Med. 2012 Jun;29(6):716-20. doi: 10.1111/j.1464-5491.2011.03547.x. PMID 22150786
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 28 centres participated: Australia (5), Germany (6), Norway (6), Sweden (5) and United States (6).
Groups:
- SIBA (D): Soluble insulin basal analogue D formulation (SIBA D, 100 dosing unit (DU)/mL (100 DU = 900 nmol), insulin degludec) was given subcutaneously once daily (OD) in the evening in combination with insulin aspart (IAsp) as meal-time insulin for 16 weeks. Insulin doses were individually adjusted.
- SIBA (E): Soluble insulin basal analogue E formulation (SIBA E, 100 dosing unit (DU)/mL (100 DU = 600 nmol), insulin degludec) was given subcutaneously once daily (OD) in the evening in combination with insulin aspart (IAsp) as meal-time insulin for 16 weeks. Insulin doses were individually adjusted.
- IGlar: Insulin glargine (IGlar) was given subcutaneously once daily (OD) in the evening in combination with insulin aspart (IAsp) as meal-time insulin for 16 weeks. Insulin doses were individually adjusted.
Period: Overall Study
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Started | 60 | 59 | 59
Exposed | 60 | 59 | 59
Completed | 55 | 52 | 52
Not Completed | 5 | 7 | 7
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Unclassified | 2 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SIBA (D) | SIBA (E) | IGlar | Total
Number analyzed (Participants) | 60 | 59 | 59 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (12.5) | 44.5 (12.7) | 47.2 (13.5) | 45.8 (12.8)
Gender [Count of Participants; unit: Participants]
  Female | 23 | 22 | 27 | 72
  Male | 37 | 37 | 32 | 106
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.5 (1.0) | 8.4 (0.9) | 8.3 (0.8) | 8.4 (0.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 10.3 (4.8) | 9.9 (3.3) | 9.5 (3.8) | 9.9 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 16 weeks of treatment
Time Frame: Week 0, Week 16
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
percentage of glycosylated haemoglobin | -0.54 (0.78) | -0.57 (0.76) | -0.62 (0.68)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG (expressed in mmol/L, 1 mg/dL = 18times mmol/L) after 16 weeks of treatment
Time Frame: Week 0, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
mmol/L | -2.06 (5.17) | -1.60 (4.66) | -0.54 (4.36)

3. Secondary Outcome: Mean of 9-point Self Measured Plasma Glucose Profile (SMPG)
Description: Estimate of the overall mean of SMPG (expressed in mmol/L, 1 mg/dL = 18times mmol/L) after 16 weeks of treatment. Plasma glucose measured: before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
mmol/L | 9.27 (0.30) | 9.56 (0.30) | 9.04 (0.30)

4. Secondary Outcome: Rate of Major and Minor Hypoglycaemic Episodes
Description: Rate of major and minor hypoglycaemic episodes per 100 patient years of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The full analysis set (FAS) included all randomised subjects.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
Episodes/100 years of patient exposure
  Major | 46 | 41 | 36
  Minor | 5838 | 5305 | 6637

5. Secondary Outcome: Rate of Nocturnal Major and Minor Hypoglycaemic Episodes
Description: Rate of nocturnal major and minor hypoglycaemic episodes per 100 patient years of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Episodes were defined as nocturnal if the time of onset was between 23:00 (included) and 06:00 (excluded).
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The full analysis set (FAS) included all randomised subjects.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
Episodes/100 years of patient exposure
  Major | 17 | 12 | 18
  Minor | 769 | 546 | 1082

6. Secondary Outcome: Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
Events/100 years of patient exposure
  Adverse events (AEs) | 653 | 874 | 914
  Serious AEs | 6 | 12 | 6
  Severe AEs | 6 | 29 | 6
  Moderate AEs | 202 | 246 | 397
  Mild AEs | 445 | 599 | 511
  Fatal AEs | 0 | 0 | 0

7. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Alanine Aminotransferase (ALAT)
Description: Laboratory values at screening (Week -1) and at Week 16
Time Frame: Week -1, Week 16
Population: The safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator. From the SAS, 55 (SIBA D), 53 (SIBA E) and 54 (IGlar) subjects contributed to the analysis at week 16.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
IU/L
  Week -1 , N=60, 59, 59 | 25.5 (11.3) | 22.7 (11.1) | 23.1 (10.2)
  Week 16 , N=55, 53, 54 | 25.0 (12.0) | 21.2 (8.0) | 23.1 (13.0)

8. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Aspartate Aminotransferase (ASAT)
Description: Laboratory values at screening (Week -1) and at Week 16
Time Frame: Week -1, Week 16
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator. From the SAS, 55 (SIBA D), 53 (SIBA E) and 54 (IGlar) subjects contributed to the analysis at week 16.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
IU/L
  Week -1, N=60, 59, 59 | 22.8 (7.4) | 21.7 (7.0) | 23.3 (11.3)
  Week 16, N=55, 53, 54 | 23.3 (8.8) | 21.6 (8.5) | 23.9 (9.4)

9. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Serum Creatinine
Description: Laboratory values at screening (Week -1) and at Week 16
Time Frame: Week -1, Week 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
umol/L
  Week -1 , N=60, 59, 59 | 77.2 (12.6) | 76.6 (12.8) | 77.6 (13.3)
  Week 16 , N=55, 53, 54 | 77.2 (14.1) | 75.9 (13.0) | 77.9 (14.5)

10. Secondary Outcome: Vital Signs: Diastolic BP (Blood Pressure)
Description: Values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator. From the SAS, 57 (SIBA E) and 57 (IGlar) subjects contributed to the analysis at week 16.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
mmHg
  Week 0 (Baseline), N=60, 59, 59 | 76 (8) | 75 (10) | 74 (9)
  Week 16, N=60, 57, 57 | 76 (10) | 75 (10) | 74 (7)

11. Secondary Outcome: Vital Signs: Systolic BP (Blood Pressure)
Description: Values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
mmHg
  Week 0 (Baseline), N=60, 59, 59 | 124 (15) | 126 (16) | 124 (16)
  Week 16, N=60, 57, 57 | 122 (14) | 125 (14) | 123 (15)

12. Secondary Outcome: Vital Signs: Pulse
Description: Values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 60 | 59 | 59
beats/minute
  Week 0 (Baseline), N=60, 59, 59 | 74 (10) | 72 (9) | 73 (10)
  Week 16, N=60, 57, 57 | 74 (12) | 72 (11) | 72 (12)

13. Secondary Outcome: Physical Examination
Description: Physical examination was performed at screening (week -1), and after 8 and 16 weeks of treatment. If any new findings or deterioration in previous findings were observed during the trial, these were recorded as AEs and are therefore not presented separately as no analysis was performed.
Time Frame: Week -1, Week 8, Week 16
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 16 weeks + 5 days follow up
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | SIBA (D) | SIBA (E) | IGlar
Serious Adverse Events (participants affected / at risk) | 1/60 | 2/59 | 1/59
Other Adverse Events (participants affected / at risk) | 31/60 | 42/59 | 31/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIBA (D) (N=60) | SIBA (E) (N=59) | IGlar (N=59)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIBA (D) (N=60) | SIBA (E) (N=59) | IGlar (N=59)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (4) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 6 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 14 (17) | 24 (29) | 15 (17)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 2 (2) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 10 (16) | 16 (35) | 10 (26)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.